CLINICAL TRIAL: NCT00003058
Title: Phase II Clinical Trial of TROGLITAZONE, a Ligand for the Peroxisome Proliferator-Activated Receptor Gamma (PPAR), as Antineoplastic Differentiation Therapy for Patients With Malignant Liposarcoma
Brief Title: Troglitazone in Treating Patients With Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, George Demetri, M.D., Demetri, George MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-075; P30CA006516 (NIH); CDR0000065717; NCI-G97-1313
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Sarcoma
Keywords: adult liposarcoma; recurrent adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Liposarcoma | interventions — Troglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Troglitazone (Experimental): Patients received troglitazone 800 mg oral once-daily. Treatment continued as long as patient was responding or in stable disease clinically and ended if patient experienced progression or unacceptable toxicity.
  Interventions: Drug: troglitazone

INTERVENTIONS:
Drug: troglitazone
  Other Names: Rezulin

SUMMARY:
Troglitazone may help liposarcoma cells develop into normal cells. This was a single arm, open-label study with a two-stage design to evaluate troglitazone in patients with liposarcoma stratified by histologic subtype.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To evaluate the clinical activity of troglitazone in patients with malignant liposarcoma stratified by histologic subtype.

II. To perform correlative imaging, biological, and biochemical testing of patients in order to define the degree to which in vivo terminal differentiation may be promoted by this therapeutic intervention.

III. To evaluate the tolerance and safety of troglitazone in this patient population.

PROJECTED ACCRUAL:

Initially, 14 patients of each of the 5 histologic subtypes of liposarcoma will be accrued. If 1 or more patients show evidence of biological response, an additional 16 patients of each subtype will be accrued for a total of 30 patients per subtype. If 4 or more of 30 patients achieve biological response then troglitazone will be deemed promising in that histologic subtype.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven liposarcoma that is incurable by standard surgery Measurable or evaluable disease required No active CNS involvement or leptomeningeal disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT less than 5 times upper normal limit Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No poorly controlled atrial arrhythmias, angina pectoris, or myocardial infarction within past 6 months No symptomatic congestive heart failure, percutaneous transluminal coronary angioplasty, or coronary artery bypass graft within past 3 months Other: Not pregnant or nursing Fertile patients must use effective contraception No known active retroviral disease

PRIOR CONCURRENT THERAPY: Recovered from toxic effects of all prior therapy No concurrent cytotoxic therapy Biologic therapy: Not specified Chemotherapy: Prior chemotherapy allowed Endocrine therapy: No concurrent hormonal therapy Radiotherapy: Prior radiation therapy for metastatic disease allowed No radiotherapy to sole site of measurable disease within past 6 months Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 1997-06; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Demetri GD, Fletcher CD, Mueller E, Sarraf P, Naujoks R, Campbell N, Spiegelman BM, Singer S. Induction of solid tumor differentiation by the peroxisome proliferator-activated receptor-gamma ligand troglitazone in patients with liposarcoma. Proc Natl Acad Sci U S A. 1999 Mar 30;96(7):3951-6. doi: 10.1073/pnas.96.7.3951. PMID 10097144
- [Result] Demetri GD, Spiegelman B, Fletcher CD, et al.: Differentiation of liposarcomas in patients treated with the PPAR g ligand troglitazone: documentation of biologic activity in myxoid/round cell and pleomorphic subtypes. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A2064, 535a, 1999.